CLINICAL TRIAL: NCT03087201
Title: A Randomized Multi-centre Double-blind Placebo Controlled Trial to Demonstrate the Efficacy and Safety of Nabiximols in the Treatment of Adults With Chronic Tic Disorders
Brief Title: CANNAbinoids in the Treatment of TICS (CANNA-TICS)
Acronym: CANNA-TICS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CANNA-TICS; 2016-000564-42 (EudraCT Number)
Record Dates: First submitted 2017-03-06; First posted 2017-03-22 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-07

CONDITIONS: Tourette Syndrome; Tic Disorders
Keywords: Chronic tic disorders; Tourette syndrome
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nabiximols, oromucosal spray (Experimental): 1-12 puffs nabiximols / day, Duration of treatment: 13 weeks
  Interventions: Drug: nabiximols
- placebo, oromucosal spray (Placebo Comparator): 1-12 puffs placebo / day, Duration of treatment: 13 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: nabiximols — starting dose (1 puff): 2.7 mg delta-9-tetrahydrocannabinol (THC) and 2.5 mg cannabidiol (CBD), maximum dose (12 puffs): 32.4 mg THC/30 mg CBD, no target dose is defined
  Duration of treatment: 13 weeks
  Arms: nabiximols, oromucosal spray
Drug: placebo — analogous to experimental intervention
  Arms: placebo, oromucosal spray

SUMMARY:
This is a multicentre, randomized, double-blind, placebo controlled, parallel-group, phase IIIb trial.

Patients (≥18 years) with chronic tic disorders and Tourette syndrome will be recruited.

The objective of the trial is to demonstrate that treatment with the cannabis extract nabiximols is superior to placebo in reducing tics and comorbidities in patients with Tourette syndrome and chronic tic disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic tic disorder or Tourette syndrome according to DSM-5
2. Age ≥18 years
3. Total tic score of the Yale Global Tic Severity Scale (YGTSS-TTS) > 14 for patients with Tourette syndrome or YGTSS-TTS > 10 for patients with chronic motor or vocal tics only (= CTD)
4. Clinical Global Impression-Severity Score (CGI-S) ≥ 4
5. Medication (and stimulation parameters for deep brain stimulation) for tics and comorbidities must be on a stable dose for at least 30 days before entering the study and patient must consent to maintain the stable dose during the study
6. Signed written informed consent and willingness to comply with treatment and follow-up procedures
7. Patients capable of understanding the investigational nature, potential risks and benefits of the clinical trial
8. Prevention of pregnancy:

Women without childbearing potential defined as follows:

* at least 6 weeks after surgical sterilization by bilateral tubal ligation or bilateral oophorectomy or
* hysterectomy or uterine agenesis or
* ≥ 50 years and in postmenopausal state ≥ 1 year or
* < 50 years and in postmenopausal state ≥ 1 year with urine FSH > 40 IU/l and urine oestrogen < 30 ng/l or a negative oestrogen test or

Women of childbearing potential with a negative urine ß-HCG pregnancy test at screening who agree to meet one of the following criteria from the time of screening, during the study and for a period of three months following the last administration of study medication:

* correct use of contraception methods. The following are acceptable: hormonal contraceptives (combined oral contraceptives, oestrogen-free pills with desogestrel, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release), intrauterine device (IUS)
* true abstinence (periodic abstinence and withdrawal are not acceptable methods of contraception)
* sexual relationship only with female partners and/or sterile male partners or Males who are not surgically sterile and who are sexually active with female partner(s) of childbearing potential must agree to correct use of one of the following contraception methods from the time of screening, during the study and for a period of three months following the last administration of study medication: hormonal contraceptives (combined oral contraceptives, oestrogen-free pills with desogestrel, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release), intrauterine device (IUS)

Exclusion Criteria:

1. Comorbid obsessive-compulsive disorder (OCD), attention deficit/hyperactivity disorder (ADHD), depression, anxiety disorder when unstable or in need of an initial adjustment for a therapy
2. Ongoing behavioural treatment for tics
3. History of schizophrenia, psychotic, severe personality, or pervasive developmental disorder
4. Patient has a history of suicidal ideation with intent to act or a plan to act in the 12 months preceding the Screening Visit
5. Current clinical diagnosis of substance abuse or dependence and compulsive disorder
6. Secondary tic disorders and other significant neurological disorders that, in the opinion of the investigator, might interfere with the patient's participation in the study, poses added risk for the patient, or confounds the assessment of patient safety
7. Severe cardiovascular diseases, hepatitis C, or other severe hepatic and renal disorders by history that, in the opinion of the investigator, might interfere with the patient's participation in the study, poses added risk for the patient, or confounds the assessment of patient safety
8. Any medical condition based on medical history, physical examination, and vital sign measurements that, in the opinion of the Investigator, might interfere with the patient's participation in the study, poses added risk for the patient, or confounds the assessment of patient safety
9. Use of cannabis or cannabinoid-based medicine (CBM) in the 30-day period prior to study entry and/or positive delta-9-tetrahydrocannabinol (THC) urine test
10. Positive urine pregnancy test
11. Pregnancy or lactation period
12. The subject has received any investigational medication or used any investigational device within 30 days prior to the first dose of study medication or is actively participating in any investigational drug or device study, or is scheduled to receive an investigational drug or to use an investigational device during the course of the study.
13. Known or suspected hypersensitivity to any of the active substances or any excipients of the investigational medicinal product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Response-rate to treatment according to YGTSS-TTS (Total Tic-Score of the Yale Global Tic Severity Scale [YGTSS]) | 13 weeks

SECONDARY OUTCOMES:
Fitness to Drive Test | 13 weeks
  Reaction time and choice reaction (RT)
Fitness to Drive Test | 13 weeks
  Stress Behavior capacity (DT-Auslastung)
Fitness to Drive Test | 13 weeks
  Stress Behavior performance quantity (DT Mengenleistung)
Fitness to Drive Test | 13 weeks
  Concentration (COG)
Fitness to Drive Test | 13 weeks
  Perceptual speed (ATAVT)
YGTSS-TTS | 8 weeks and 1 month after end of treatment (17 weeks)
YGTSS-TTS | Baseline and 13 weeks
YGTSS-Global Score (YGTSS-GS) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)
Modified Rush Video-Based Tic Rating Scale (MRVS) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)
Clinical Global Impression-Improvement Score (CGI-I) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)
Clinical Global Impression-Severity Score (CGI-S) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)
Adult Tic Questionnaire (ATQ) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)
Tourette Syndrome-Quality of Life Scale (GTS-QoL) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)
Pre-monitory Urge for Tics Scale (PUTS) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)
Beck Depression Inventory-II (BDI-II) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)
Conners' Adult ADHD Rating Scale (CAARS) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)
Beck Anxiety Inventory (BAI) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)
Pittsburgh Sleep Quality Index (PSQI) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)
Skala Impulsives-Verhalten-8 (I-8) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)
12-item short-form Health Survey (SF-12) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)
Rage Attacks Questionnaire for Adults with GTS (RAQ-GTS) | 8 weeks, 13 weeks and 1 month after end of treatment (17 weeks)

OTHER OUTCOMES:
Assessment of adverse events (AEs) | through study completion, an average of 17 weeks
Assessment of serious adverse events (SAEs) | through study completion, an average of 17 weeks
blood pressure | through study completion, an average of 17 weeks
pulse | through study completion, an average of 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Müller-Vahl, MD, Principal Investigator — Hannover Medical School, Clinic of Psychiatry, Socialpsychiatry and Psychotherapy
Locations (6):
- Germany (6):
  - Uniklinik RWTH Aachen, Psychiatry and Psychotherapy, Aachen
  - University Hospital Cologne, Psychiatry and Psychotherapy, Cologne
  - University of Freiburg, Psychiatry and Psychotherapy, Freiburg im Breisgau
  - Hannover Medical School, Clinic of Psychiatry, Socialpsychiatry and Psychotherapy, Hanover
  - University Hospital Schleswig-Holstein, Institute of Neurogenetics, Department of Pediatric and Adult Movement Disorders and Neuropsychiatrics, Lübeck
  - LMU Munich, Psychiatry and Psychotherapy, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szejko N, Saramak K, Lombroso A, Muller-Vahl K. Cannabis-based medicine in treatment of patients with Gilles de la Tourette syndrome. Neurol Neurochir Pol. 2022;56(1):28-38. doi: 10.5603/PJNNS.a2021.0081. Epub 2021 Oct 28. PMID 34708399
- [Derived] Jakubovski E, Pisarenko A, Fremer C, Haas M, May M, Schumacher C, Schindler C, Hackl S, Aguirre Davila L, Koch A, Brunnauer A, Cimpianu CL, Lutz B, Bindila L, Muller-Vahl K. The CANNA-TICS Study Protocol: A Randomized Multi-Center Double-Blind Placebo Controlled Trial to Demonstrate the Efficacy and Safety of Nabiximols in the Treatment of Adults With Chronic Tic Disorders. Front Psychiatry. 2020 Nov 26;11:575826. doi: 10.3389/fpsyt.2020.575826. eCollection 2020. PMID 33324255